CLINICAL TRIAL: NCT02098161
Title: Open Label Phase 2 Single Agent Study of LCL-161 in Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (Post-PV MF), or Post-Essential Thrombocytosis Myelofibrosis (Post-ET MF)
Brief Title: LCL161 in Treating Patients With Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocytosis Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0612; NCI-2014-01241 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CLCL161AUS02T; 2013-0612 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Primary Myelofibrosis | interventions — LCL161

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SMAC mimetic LCL161) (Experimental): Patients receive SMAC mimetic LCL161 PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Drug: Smac Mimetic LCL161

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Drug: Smac Mimetic LCL161 — Given PO
  Other Names: LCL161

SUMMARY:
This phase II trial studies how well second mitochondrial-derived activator of caspases (SMAC) mimetic LCL161 (LCL161) works in treating patients with primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocytosis myelofibrosis. SMAC mimetic LCL161 may help control the growth of abnormal cells by promoting apoptosis (programmed cell death).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of LCL161 as therapy for primary myelofibrosis (PMF), post-polycythemia vera (PV) myelofibrosis (MF) and post-essential thrombocytosis (ET) MF.

II. To determine the objective response which is defined as CR (complete remission) + PR (partial remission) + CI (clinical improvement) after three cycles of treatment.

SECONDARY OBJECTIVES:

I. To determine the safety of LCL161 as therapy for PMF, post-PV MF and post-ET MF.

II. To determine time to response and response duration. III. To assess changes in symptom burden as assessed by Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) and M.D. Anderson Symptom Inventory (MDASI) questionnaires.

EXPLORATORY OBJECTIVE:

I. To assess the mechanisms of action of LCL161 in patients with MF; these studies will include the analysis of baculoviral IAP repeat containing 2 (cIAP1), X-linked inhibitor of apoptosis, E3 ubiquitin protein ligase (XIAP), and poly (adenosine diphosphate [ADP]-ribose) polymerase 1 (PARP) protein levels which will be determined by western blot (actin as loading control) and will be measured at baseline and at beginning of each cycle for first 3 cycles and at end of study.

OUTLINE:

Patients receive SMAC mimetic LCL161 orally (PO) on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Patient is able to swallow and retain oral medication
* Must be diagnosed with treatment requiring PMF or post ET/PV MF with intermediate-1, intermediate -2 or high risk disease according to the International Working Group (IWG) prognostic scoring system, or if with low risk disease then with symptomatic splenomegaly that is >= 5 cm below left costal margin by physical exam
* Patients who are not candidates for, intolerant, or relapsed/refractory to ruxolitinib
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 0.5 x 10^9/L (1500/mm^3)
* Serum direct bilirubin =< 2.0 x ULN (upper limit of normal)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN, except for patients with MF involvement of the liver who must have AST and ALT =< 5 x ULN
* Serum creatinine =< 1.5 x ULN
* Treatment-related toxicities from prior therapies must have resolved to grade =< 1
* At least 2 weeks from prior MF-directed treatment (till the start of study drug)

Exclusion Criteria:

* Any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while in the study or that could confound discrimination between disease- and study treatment-related toxicities
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following: history or presence of ventricular tachyarrhythmia; presence of unstable atrial fibrillation (ventricular response > 100 beats per minute [bpm]); patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria; clinically significant resting bradycardia (< 50 bpm); angina pectoris or acute myocardial infarction =< 3 months prior to starting study drug; other clinically significant heart disease (e.g., symptomatic congestive heart failure; uncontrolled arrhythmia or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen)
* Patients who are currently receiving chronic (> 14 days) treatment with corticosteroids at a dose >= 10 mg of prednisone (or its glucocorticoid equivalent) per day, or any other chronic immunosuppressive treatment that cannot be discontinued prior to starting study drug
* Patients who are currently receiving treatment with agents that are metabolized solely through cytochrome P450 family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) and have a narrow therapeutic index or are strong cytochrome P450 family 3, subfamily C, polypeptide 8 (CYP2C8) inhibitors; or are receiving treatment with agents that carry a risk for QT prolongation and are CYP3A substrates
* Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LCL161 as per physicians opinion
* Pregnant or breast feeding (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive beta-human chorionic gonadotropin (HCG) laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 90 days after study treatment; highly effective contraception methods include: total abstinence or male partner or female sterilization or combination of any two of the following (a+b or a+c, or b+c): a) use of oral, injected or implanted hormonal methods of contraception, b) placement of an intrauterine device (IUD) or intrauterine system (IUS), c) barrier methods of contraception: condom for male partner or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

  * Note: postmenopausal women are allowed to participate in this study; women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, a woman is considered to be of not child bearing potential only when her reproductive status has been confirmed by follow-up hormone level assessment
* Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping study drug and should not father a child in this period; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pemmaraju, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pemmaraju N, Carter BZ, Bose P, Jain N, Kadia TM, Garcia-Manero G, Bueso-Ramos CE, DiNardo CD, Bledsoe S, Daver NG, Popat U, Konopleva MY, Zhou L, Pierce S, Estrov ZE, Borthakur GM, Ohanian M, Qiao W, Masarova L, Wang X, Mak PY, Cortes J, Jabbour E, Verstovsek S. Final results of a phase 2 clinical trial of LCL161, an oral SMAC mimetic for patients with myelofibrosis. Blood Adv. 2021 Aug 24;5(16):3163-3173. doi: 10.1182/bloodadvances.2020003829. PMID 34424319
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (SMAC Mimetic LCL161)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (SMAC Mimetic LCL161)
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 37
Age, Continuous [Median (Full Range); unit: years] | 72 [56 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 42
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Will be defined as complete remission (CR), partial remission (PR), or clinical improvement (CI) after 3 courses of treatment according to International Working Group (IWG) consensus criteria for myelofibrosis. Complete remission (CR): bone marrow blasts <5%, hemoglobin >/= 10, absolute neutrophil count (ANC) >/= 1000, platelets >/= 100, <2% immature myeloid cell, spleen and liver not palpable. Partial Response (PR): CR plus one or more of the following: ANC >/= 1000, decreased platelets by 50%, hemoglobin >/= 8.5 but < 10, <2% immature myeloid cells. Clinical improvement (CI): hemoglobin increase of 2g/dl, transfusion independence or reduction splenomegaly and/or hepatomegaly >/= 50%, >/=50% reduction in MPN-SAF TSS
Time Frame: After 3 courses of Therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SMAC Mimetic LCL161)
Number analyzed (Participants) | 50
Participants | 15

2. Secondary Outcome: Duration of Response
Description: duration of response is defined as the date at which the subject's objective status is first noted to be a CR or PR to the date progression is documented (if one has occurred) or to the date of last follow-up (for those subjects who have not progressed).
Time Frame: Up to 7 years 5 Months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (SMAC Mimetic LCL161)
Number analyzed (Participants) | 50
Months | 31.5 [3.6 to 59.2]

3. Secondary Outcome: Time to Response
Description: The time to response is defined as the time from study registration to the first date at which the subject's objective status was classified as a response (CR or PR). In subjects who do not achieve a response, time to response will be censored at the subject's last evaluation date. The distribution for each of these event-time variables (duration of response and time to response) will be estimated by Kaplan-Meier curves.
Time Frame: Up to 7 years 5 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (SMAC Mimetic LCL161)
Number analyzed (Participants) | 50
Months | 1.4 [0.9 to 9.1]

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 7 years 5 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (SMAC Mimetic LCL161)
Number analyzed (Participants) | 50
Months | 34 [2.2 to 60.1]

ADVERSE EVENTS:
Time Frame: Up to 7 years 5 months
Arm/Group | Treatment (SMAC Mimetic LCL161)
All-Cause Mortality (participants affected / at risk) | 2/50
Serious Adverse Events (participants affected / at risk) | 33/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SMAC Mimetic LCL161) (N=50)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 (3)
Chest pain cardiac (Cardiac disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 5 (5)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Lung infection (Infections and infestations) | 9 (11)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6)
Nervous system disorders (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Sepsis (Infections and infestations) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2)
Syncope (Nervous system disorders) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SMAC Mimetic LCL161) (N=50)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 3 (3)
Confusion (Psychiatric disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Flushing (Vascular disorders) | 3 (3)
Gait disturbance (General disorders) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Lightheadedness (Nervous system disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (4)
Memory impairment (Nervous system disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Malaise (General disorders) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Flu like symptoms (General disorders) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Urinary frequency (Renal and urinary disorders) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Bruising (Injury, poisoning and procedural complications) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Chills (General disorders) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 8 (9)
Hypotension (Vascular disorders) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9)
night sweats (General disorders) | 7 (9)
Insomnia (Psychiatric disorders) | 8 (10)
Weight loss (Investigations) | 10 (10)
Constipation (Gastrointestinal disorders) | 12 (12)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 (13)
Surgical and medical procedures (Surgical and medical procedures) | 6 (13)
Fever (General disorders) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14)
Abdominal distension (Gastrointestinal disorders) | 15 (15)
Headache (General disorders) | 15 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (22)
Edema limbs (General disorders) | 19 (20)
Investigations (Investigations) | 8 (20)
Vomiting (Gastrointestinal disorders) | 20 (20)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 21 (21)
Dizziness (Nervous system disorders) | 23 (23)
Infection (Infections and infestations) | 15 (23)
Diarrhea (Gastrointestinal disorders) | 27 (27)
Pain (General disorders) | 33 (60)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (28)
Nausea (Gastrointestinal disorders) | 35 (35)
Fatigue (General disorders) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT02098161/Prot_SAP_000.pdf